CLINICAL TRIAL: NCT00751634
Title: Temperature Control in Central Fever in the Neuro-ICU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Gaymar Industries, Inc. (Industry)
Responsible Party: Principal Investigator, Andrew Naidech, Associate Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1507-009
Record Dates: First submitted 2008-09-10; First posted 2008-09-12 (Estimated); Results first posted 2012-04-09 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-04

CONDITIONS: Fever; Brain Hemorrhage
Keywords: subarachnoid hemorrhage; intracerebral hemorrhage; fever
MeSH Terms: conditions — Fever; Intracranial Hemorrhages; Subarachnoid Hemorrhage; Cerebral Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Application of the Gaymar Rapr-Round device per approved use
  Interventions: Device: Gaymar Rapr-Round (external cooling blanket)

INTERVENTIONS:
Device: Gaymar Rapr-Round (external cooling blanket) — Application of the device per its approved labeling

SUMMARY:
There are few treatments for central fever (fever that is due to the central nervous system, as opposed to an infectious source). We hypothesize that an externally applied cooling blanket will reduce temperature in neurologically ill patients with central fever.

ELIGIBILITY:
Inclusion Criteria:

* Two or more days with core temperature ≥ 100.4F
* Approval of the patient's primary attending physician
* Need for core temperature measurement independent of the study.
* Admission to the Neuro-ICU [intensive care unit] for an underlying condition

Exclusion Criteria:

* Evidence for an infectious cause of fever, such as pneumonia, bacteremia, CNS [central nervous system] infection or urinary tract infection.
* Expected death from any cause
* Known sensitivity to the device
* History of pre-admission hypothalamic dysfunction or known temperature dysregulation
* Use of 2 or more vasopressor medications, since this may make a local skin reaction to the device more likely
* Hemodynamic instability

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Naidech, MD MSPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: Application of the Gaymar Rapr-Round device per FDA-approved use (temperature reduction in patients with fever in a monitored setting)
Period: Overall Study
Arm/Group | Treatment Group
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 54.3 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Core Temperature as Measured With an Approved Device (Urinary Catheter) in Place for Usual Clinical Care
Description: Core temperature (in degrees Fahrenheit, F) throughout the study period. The cooling blanket was in place throughout the study period unless severe shivering led to termination per protocol.
Time Frame: baseline, one, two and six hours after application.
Measure: Mean (Standard Deviation); unit: degrees F
Groups:
- Treatment Group at 0, 1, 2, 6 Hours: Application of the Gaymar Rapr-Round device per approved use
Arm/Group | Treatment Group at 0, 1, 2, 6 Hours
Number analyzed (Participants) | 20
degrees F
  0 hours | 100.8 (0.4)
  1 hour | 100.3 (0.9)
  2 hours | 99.9 (1.1)
  6 hours | 99.5 (0.7)

2. Secondary Outcome: Time From Start of Cooling Device to Core Temperature < 100.4F
Description: For all patients, the time until the core temperature (measured with a urinary catheter in place for usual clinical care) was <100.4F
Time Frame: Six hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment Group
Number analyzed (Participants) | 20
hours | 2.1 (1.6)

3. Secondary Outcome: Number of Participants With Severe Shivering
Description: Severe shivering as measured by the bedside shivering assessment scale: 0 None: no shivering noted on palpation of the masseter, neck, or chest wall
  1. Mild: shivering localized to the neck and/or thorax only
  2. Moderate: shivering involves gross movement of the upper extremities (in addition to neck and thorax)
  3. Severe: shivering involves gross movements of the trunk and upper and lower extremities
Time Frame: six hours
Population: All participants were analyzed for the outcome of BSAS=3
Measure: Number; unit: participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 20
participants | 4

4. Secondary Outcome: Number of Participants With Hypotension
Description: New systolic blood pressure < 100 mm Hg, or new vasopressor use during study period
Time Frame: six hours
Measure: Number; unit: participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 20
participants | 0

5. Secondary Outcome: Number of Participants With Arrhythmia
Description: New ventricular tachycardia, ventricular fibrillation, atrial fibrillation or other unstable cardiac rhythm
Time Frame: Six hours
Measure: Number; unit: participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 20
participants | 0

ADVERSE EVENTS:
Arm/Group | Treatment Group
Serious Adverse Events (participants affected / at risk) | 4/20
Other Adverse Events (participants affected / at risk) | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=20)
Shivering (Nervous system disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days